CLINICAL TRIAL: NCT01651442
Title: Sequenced Therapies for Comorbid and Primary Insomnias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jack Edinger, PhD (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Jack Edinger, PhD, Principal Investigator, National Jewish Health
Organization: National Jewish Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH091053-01 (NIH); R01MH091075 (NIH)
Record Dates: First submitted 2012-06-26; First posted 2012-07-27 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2019-08

CONDITIONS: Insomnia Comorbid to Psychiatric Disorder; Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; Trazodone; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Non-drug Sleep Therapy 1 (Active Comparator)
  Interventions: Behavioral: Behavioral Insomnia Therapy
- Sleep Medication 1 (Active Comparator)
  Interventions: Drug: Zolpidem
- Non-drug Sleep Therapy 2 Following Non-drug Sleep Therapy 1 (Active Comparator)
  Interventions: Behavioral: Cognitive Therapy
- Sleep Medication 2 Following Sleep Medication 1 (Active Comparator)
  Interventions: Drug: Trazodone
- Non-drug Sleep Therapy 1 Following Sleep Medication 1 (Active Comparator)
  Interventions: Behavioral: Behavioral Insomnia Therapy
- Sleep Medication 1 Following Non-drug Sleep Therapy 1 (Active Comparator)
  Interventions: Drug: Zolpidem

INTERVENTIONS:
Behavioral: Behavioral Insomnia Therapy — Sleep hygiene, stimulus control, and sleep restriction presented in four sessions.
  Arms: Non-drug Sleep Therapy 1; Non-drug Sleep Therapy 1 Following Sleep Medication 1
Drug: Zolpidem — 5mg or 10mg
  Arms: Sleep Medication 1; Sleep Medication 1 Following Non-drug Sleep Therapy 1
Drug: Trazodone — 50mg to 150mg
  Arms: Sleep Medication 2 Following Sleep Medication 1
Behavioral: Cognitive Therapy — Cognitive restructuring, constructive worry, behavioral experiments presented in four sessions.
  Arms: Non-drug Sleep Therapy 2 Following Non-drug Sleep Therapy 1

SUMMARY:
Chronic insomnia is a prevalent disorder associated with increased health care costs, impaired functioning, and an increased risk for developing serious psychiatric disorders. Cognitive-behavioral therapies (CBTs) and benzodiazepine receptor agonist (BzRA) medications are the most widely supported approaches for insomnia management. Unfortunately, few studies have compared the psychological/behavioral therapies and BzRAs for insomnia treatment. Moreover, insomnia treatment studies have been limited by small, highly screened study samples, fixed-dose and fixed-agent pharmacotherapy strategies that do not represent usual adjustable dosing practices, relatively short follow-up intervals, and reliance on self-report or polysomnographic (PSG) sleep parameters as outcomes, rather than on more clinically relevant indicators of remission. Finally, studies have yet to test the benefits of treatment sequencing for those who do not respond to initial their insomnia therapy. This multi-site project will address these limitations. Two study sites will enroll a total of 224 participants who meet broad criteria for a chronic insomnia disorder, and a sizeable portion (60%) of this sample will have insomnia occurring comorbid to a psychiatric disorder. Participants will be evaluated with clinical assessments and PSG, and then will be randomly assigned to first-stage therapy with an easy-to-administer behavioral insomnia therapy (BT) or zolpidem (most widely prescribed BzRA). Centrally trained therapists will administer therapies according to manualized, albeit flexible, treatment algorithms. Initial outcomes will be assessed after 6 weeks, and treatment remitters will be followed for the next 12 months on maintenance therapy. Those not achieving remission will be offered re-randomization to a second, 6-week treatment involving pharmacotherapy (zolpidem or trazodone) or psychological therapy (BT or cognitive therapy-CT). All participants will be re-evaluated 12 weeks after protocol initiation, and at 3-, 6-, 9-, and 12-month follow-ups while continuing their final treatment. Insomnia remission, defined categorically as a score < 8 on the Insomnia Severity Index, will serve as the primary outcome for treatment comparisons. Secondary outcomes will include sleep diary and PSG sleep measures; subjective ratings of sleep and daytime function; adverse events; dropout rates; and treatment acceptability. Our over-arching goal is to obtain new information that aids in the development of clinical guidelines for managing insomnia sufferers with and without comorbid psychiatric conditions.

ELIGIBILITY:
Inclusion Criteria:

* a complaint of persistent (i.e., > 1 month) difficulties initiating or maintaining sleep despite adequate opportunity for sleep;
* a sleep onset latency or wake time after sleep onset > 30 minutes 3 or more nights per week during two weeks sleep diary monitoring;
* an Insomnia Severity Index (ISI) score > 10 indicating at least "mild" insomnia; and
* a score ≥ 2 on either the interference or distress item of the screening ISI, indicating the insomnia causes significant distress or impairment in social, occupational, or other areas of functioning. These criteria represent those provided in the DSM-IV-TR87, Research Diagnostic Criteria3 and the International Classification of Sleep Disorders4, and will ensure a sample with clinically relevant insomnia.

Exclusion Criteria:

Exclusion criteria will be minimal to retain a broadly representative sample that includes patients with primary and insomnia comorbid to a psychiatric disorder. Likewise, individuals with a comorbid medical condition will be excluded only if the medical condition is life-threatening or would contra-indicate using study medications. Exclusion criteria are

* an untreated psychiatric disorder (e.g., major depression) as these conditions have specific treatments and it would be inappropriate not to offer those treatments;
* a lifetime diagnosis of any psychotic or bipolar disorder as sleep restriction and medications for insomnia may precipitate mania and hallucinations;
* an imminent risk for suicide;
* alcohol or drug abuse within the past year, since BzRAs are cross-tolerant with alcohol;
* terminal or progressive physical illness (e.g., cancer, COPD), or neurological degenerative disease (e.g., dementia);
* current use of medications known to cause insomnia (e.g., steroids);
* sleep apnea (apnea/hypopnea index > 15), restless legs syndrome, periodic limb movement during sleep (PLMS with arousal > 15 per hour), or a circadian rhythm sleep disorder (e.g., advanced sleep phase syndrome);
* habitual bedtimes later than 2:00 AM or rising times later than 10:00 AM;
* consuming > 2 alcoholic beverages per day on a regular basis.

Individuals using sleep-aids (prescribed or over-the-counter) will be included if they are willing and able to discontinue medications at least 2 weeks before baseline assessment. Participants using alcohol as a sleep aid or alcohol after 7:00pm on a regular basis will be required to discontinue this practice at least two weeks prior to baseline assessment. Individuals using psychotropic medications (e.g., anxiolytics, antidepressants) will not be automatically excluded from the study. Those on stable dosages (for at least three months) of SSRI or SNRI medications and who show at least partial remission (via SCID) from their mood or anxiety disorder will be accepted in the study if they meet the selection criteria above. Patients using TCAs, MAOIs, or atypical antidepressants will be excluded even if in remission as the effects of these medications on sleep might confound interpretation of the findings. We will impose similar standards for those with MDD, dysthymia, panic disorder, phobia, and GAD. We realize that some decisions about enrollment may not always be easy to make, but we will rely on all available data and a consensus approach to guide our clinical decision making process

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Edinger, PhD, Principal Investigator — National Jewish Health; Charles Morin, PhD, Principal Investigator — Universite Laval
Locations (2):
- National Jewish Health, Denver, Colorado, United States
- Université Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Morin CM, Chen SJ, Ivers H, Beaulieu-Bonneau S, Krystal AD, Guay B, Belanger L, Cartwright A, Simmons B, Lamy M, Busby M, Edinger JD. Effect of Psychological and Medication Therapies for Insomnia on Daytime Functions: A Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2349638. doi: 10.1001/jamanetworkopen.2023.49638. PMID 38153735
- [Derived] Edinger JD, Beaulieu-Bonneau S, Ivers H, Guay B, Belanger L, Simmons B, Morin CM. Association between insomnia patients' pre-treatment characteristics and their responses to distinctive treatment sequences. Sleep. 2022 Jan 11;45(1):zsab245. doi: 10.1093/sleep/zsab245. PMID 34792177
- [Derived] Morin CM, Edinger JD, Beaulieu-Bonneau S, Ivers H, Krystal AD, Guay B, Belanger L, Cartwright A, Simmons B, Lamy M, Busby M. Effectiveness of Sequential Psychological and Medication Therapies for Insomnia Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Nov 1;77(11):1107-1115. doi: 10.1001/jamapsychiatry.2020.1767. PMID 32639561
- [Derived] Morin CM, Edinger JD, Krystal AD, Buysse DJ, Beaulieu-Bonneau S, Ivers H. Sequential psychological and pharmacological therapies for comorbid and primary insomnia: study protocol for a randomized controlled trial. Trials. 2016 Mar 3;17(1):118. doi: 10.1186/s13063-016-1242-3. PMID 26940892

RESULTS

PARTICIPANT FLOW:
Period: Phase I Treatment
Arm/Group | Non-drug Sleep Therapy 1 | Sleep Medication 1 | Non-drug Sleep Therapy 2 Following Non-drug Sleep Therapy 1 | Sleep Medication 2 Following Sleep Medication 1 | Non-drug Sleep Therapy 1 Following Sleep Medication 1 | Sleep Medication 1 Following Non-drug Sleep Therapy 1
Started | 104 | 107 | 0 | 0 | 0 | 0
Completed | 88 | 80 | 0 | 0 | 0 | 0
Not Completed | 16 | 27 | 0 | 0 | 0 | 0
Period: Phase II Treatment
Arm/Group | Non-drug Sleep Therapy 1 | Sleep Medication 1 | Non-drug Sleep Therapy 2 Following Non-drug Sleep Therapy 1 | Sleep Medication 2 Following Sleep Medication 1 | Non-drug Sleep Therapy 1 Following Sleep Medication 1 | Sleep Medication 1 Following Non-drug Sleep Therapy 1
Started | 0 | 0 | 27 | 27 | 27 | 27
Completed | 0 | 0 | 25 | 15 | 21 | 17
Not Completed | 0 | 0 | 2 | 12 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-drug Sleep Therapy 1 | Sleep Medication 1 | Total
Number analyzed (Participants) | 104 | 107 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.4) | 45.4 (15.5) | 45.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 68 | 132
  Male | 40 | 39 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 94 | 93 | 187
  Black | 6 | 8 | 14
  Other | 3 | 3 | 6
  Hispanic | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Met Remission as Measured by the Insomnia Severity Index
Description: The Insomnia Severity Index (ISI) is a self-report questionnaire assessing the nature, severity, and impact of insomnia. Remission is determined to be a score less-than 8.
Time Frame: 6 weeks, 12 weeks, 3 months, 6 months, 9 months & 12 months
Measure: Number; unit: percent remitted
Groups:
- Sleep Medication 1 Plus Non-drug Sleep Therapy 1: Zolpidem Plus Behavioral Therapy
- Sleep Medication 1 Plus Sleep Medication 2: Zolpidem Plus Trazodone
- Non-drug Sleep Therapy 1 Plus Non-drug Sleep Therapy 1: Behavioral Therapy Plus Cognitive Therapy
- Non-drug Sleep Therapy 1 Plus Sleep Medication 1: Behavioral Therapy Plus Zolpidem
Arm/Group | Non-drug Sleep Therapy 1 | Sleep Medication 1 | Sleep Medication 1 Plus Non-drug Sleep Therapy 1 | Sleep Medication 1 Plus Sleep Medication 2 | Non-drug Sleep Therapy 1 Plus Non-drug Sleep Therapy 1 | Non-drug Sleep Therapy 1 Plus Sleep Medication 1
Number analyzed (Participants) | 90 | 83 | 27 | 27 | 27 | 27
percent remitted | 40.00 | 34.94 | 37.04 | 48.15 | 44.44 | 55.56

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the period from March 1, 2012 to July 1, 2017. Adverse Events were monitored in participants during the entirety of their participation, up to approximately 17 months for each participant.
Groups:
- Non-drug Sleep Therapy 2: Cognitive Therapy: Cognitive restructuring, constructive worry, behavioral experiments presented in four sessions.
- Sleep Medication 2: Trazodone: 50mg to 150mg
Arm/Group | Non-drug Sleep Therapy 1 | Sleep Medication 1 | Non-drug Sleep Therapy 2 | Sleep Medication 2
All-Cause Mortality (participants affected / at risk) | 0/131 | 0/134 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/131 | 0/134 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/131 | 0/134 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT01651442/Prot_SAP_000.pdf